CLINICAL TRIAL: NCT05237362
Title: An Effectiveness-implementation Hybrid Trial to Evaluate a Health Promotion Intervention Within Swedish Primary Child Healthcare: Saga Stories in Health Talks
Brief Title: Saga Stories in Health Talks in Primary Child Healthcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Marie Löf, docent, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-06106-01
Record Dates: First submitted 2022-01-21; First posted 2022-02-14 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Self Efficacy
Keywords: Health promotion; Primary child healthcare

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receives the Saga Stories health promotion talk as well as take-home material
  Interventions: Behavioral: Saga Stories
- Control (No Intervention): Receives standard health promotion talk

INTERVENTIONS:
Behavioral: Saga Stories — Saga Stories in health talks consists of material for child healthcare nurses to use to facilitate the health talk with both the child and parent(s) and is complemented with take-home material. Every nurse will receive a large flip-chart with colourful pictures and text to facilitate their health talk at the 5-year check-up. The flip-chart will include information and questions regarding food, physical activity and sedentary behaviour, sleep, dental health, as well as bathroom habits. At the conclusion of the check-up the children will receive the book 'Saga Stories: Your amazing body and brain´ as well as games for the child to take home to promote healthy lifestyle behaviours (fruit and vegetable bingo and a physical activity fortune teller).
  Arms: Intervention

SUMMARY:
Primary child healthcare in Sweden is an important arena for health promotion interventions as nurses regularly meet parents and children from birth to five years of age. To date there is a lack of evidence-based material for child healthcare nurses to use in health promotion talks within primary child healthcare. Therefore, the aims of this study are to: (i) evaluate the effectiveness of Saga Stories in health talks on parental self-efficacy to promote healthy diet, physical activity, and screen time behaviours in 5-year-old children and (ii) evaluate the implementation of Saga Stories in health talks with regards to acceptability, appropriateness, feasibility, fidelity, adoption, sustainability, satisfaction, and usage.

ELIGIBILITY:
Inclusion Criteria:

* The parent the accompanies the child to the 5-year check-up at primary child healthcare needs to be able to understand Swedish sufficiently well in order to provide informed consent and partake in the Saga Stories health talk.

Exclusion Criteria:

* None

Ages: 5 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 763 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Self-efficacy | At the end of the intervention which is two months after baseline
  Parental self-efficacy for promoting healthy dietary and physical activity behaviours in their children´ questionnaire

SECONDARY OUTCOMES:
Intake of key dietary indicators as assessed by a questionnaire | At the end of the intervention which is two months after baseline
  Intake of fruits, vegetables, and sugar sweetened drinks (grams/day)
Screen time as assessed by a questionnaire | At the end of the intervention which is two months after baseline
  Number of minutes per day spent in front of a screen
Acceptability | 3 months after implementation
  Acceptability of the Saga Stories intervention by the child healthcare nurses (assessed by the questionnaire by Weiner et al.) It includes four questions assessed on a five point likert scale ranging from completely disagree to completely agree.
Appropriateness | 3 months after implementation
  Appropriateness of the Saga Stories intervention by the child healthcare nurses (assessed by the questionnaire by Weiner et al.) It includes four questions rated on a five point likert scale ranging from completely disagree to completely agree.
Feasibility of implementing Saga Stories | 3 months after implementation
  Feasibility of the Saga Stories intervention by the child healthcare nurses (assessed with by questionnaire by Weiner et al.) It includes four questions rated on a five point likert scale ranging from completely disagree to completely agree.
Change in the fidelity of the Saga Stories intervention | 2, 4, 6, 8, 10, and 12 months after implementation
  Assessment based on checklist developed for this study (0, not implemented and 1, implemented)
Change in the adoption of the Saga Stories intervention | 2, 4, 6, 8, 10, and 12 months after implementation
  Assessment based on checklist developed for this study (0, not implemented and 1, implemented)
Sustainability | One year after implementation
  Semi-structured interviews with primary child healthcare nurses
Parental satisfaction and usage of Saga Stories | Post-intervention (i.e., 2 months after baseline assessment)
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biosciences and Nutrition, Karolinska Institutet, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henstrom M, Delisle Nystrom C, Andermo S, Thomas K, Lof M. 'Saga Stories in health talks' for health promotion in Swedish child healthcare: results from a cluster-randomised hybrid type 1 effectiveness-implementation study. BMC Public Health. 2025 May 2;25(1):1637. doi: 10.1186/s12889-025-22786-1. PMID 40316984
- [Derived] Delisle Nystrom C, Henstrom M, Andermo S, Almquist-Tangen G, Thomas K, Lof M. Study protocol for an effectiveness-implementation hybrid trial to evaluate a health promotion intervention in parents and their 5-year-old child: Saga Stories in health talks in Swedish child healthcare. BMC Public Health. 2022 Nov 25;22(1):2184. doi: 10.1186/s12889-022-14549-z. PMID 36434605